CLINICAL TRIAL: NCT01561950
Title: Use of Recombinant FVIIa to Mitigate Clopidogrel Anti-platelet Therapy-Mediated Bleeding in a Single Centre, Randomized, Placebo-controlled, Double-blind Clinical Trial
Brief Title: Efficacy of Activated Recombinant Human Factor VII in Healthy Volunteers Treated for Punch Biopsy Mediated Bleeding
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F7HAEM-1955
Record Dates: First submitted 2012-03-21; First posted 2012-03-23 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Haemostasis; Healthy
MeSH Terms: interventions — Factor VII; Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Factor VII (Experimental)
  Interventions: Drug: eptacog alfa (activated); Drug: clopidogrel
- Placebo (Placebo Comparator)
  Interventions: Drug: clopidogrel; Drug: placebo

INTERVENTIONS:
Drug: eptacog alfa (activated) — If subject is eligible to continue after clopidogrel treatment, three different doses of trial drug is administered i.v. as a slow bolus injection over two to three minutes followed by post-trial biopsies
  Other Names: activated recombinant human factor VII
  Arms: Factor VII
Drug: clopidogrel — Following a baseline biopsy (B0) subjects will receive oral treatment with an initial 300 mg loading dose followed by daily 75 mg doses for at least 3 additional days. If the target platelet inhibition (PI) is achieved, the subject will undergo punch biopsy 1 (B1).
Drug: placebo — If subject is eligible to continue after clopidogrel treatment, three different doses of trial drug is administered i.v. as a slow bolus injection over two to three minutes followed by post-trial biopsies
  Arms: Placebo

SUMMARY:
This trial is conducted in the United States of the America (USA). The aim of this trial is to evaluate the effectiveness of activated recombinant human factor VII to mitigate experimentally-induced bleeding in healthy volunteers treated with clopidogrel (Plavix®).

ELIGIBILITY:
Inclusion Criteria:

* PT/PTT within normal laboratory range (e.g., PT: 9.4-12.0)
* Platelet count within normal laboratory range

Exclusion Criteria:

* The receipt of any investigational drug within 1 month prior to this trial
* Use of anticoagulation therapy-defined as vitamin K antagonists, platelet antagonists, heparin
* (or low molecular weight heparin), aspirin or NSAIDs (non-steroidal anti-inflammatory drug) within 30 days prior to trial
* African-American race
* Weight above or equal to 160 kg

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2008-05; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Bleeding duration measured in minutes | From onset of bleeding till the end of the bleeding

SECONDARY OUTCOMES:
Blood volume reported in millilitres | From onset of bleeding till the end of the bleeding
Clot dynamics on the TEG (thromboelastograph hemostasis analyzer): R in minutes | Time to onset of clot formation
Clot dynamics on the TEG (thromboelastograph hemostasis analyzer): K in minutes | Time to achieve 20 mm clot strength
Adverse events, including thrombotic events | From screening to day 11-18
Change in coagulation-related parameters after pre-biopsy | From baseline to 15 minutes after pre-biopsy
Change in coagulation-related parameters after biopsy B2 | From baseline to 3 hours after B2
Change in coagulation-related parameters after biopsy B3 | From baseline to 1 hour after B3

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neptune City, New Jersey, United States

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com